CLINICAL TRIAL: NCT04844775
Title: EHVA P01/ANRS VRI08: A Prophylactic HIV Vaccine Trial to Evaluate the Safety and Immunogenicity of HIV Clade C DREP Alone and in Combination With a Clade C ENV Protein in Healthy HIV-uninfected Adults
Brief Title: A Prophylactic HIV Vaccine Trial to Evaluate the Safety and Immunogenicity of HIV Clade C DREP Alone and in Combination With a Clade C ENV Protein in Healthy HIV-uninfected Adults
Acronym: EHVA P01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Medical Research Council (Other Government); Henri Mondor University Hospital (Other); Chelsea and Westminster Hospital, UK (Unknown); EuroVacc Foundation (Other); European Commission (Other); Swiss Government (Unknown); University College London Hospitals (Other); Imperial College London (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EHVA P01/ANRS VRI08
Record Dates: First submitted 2021-03-24; First posted 2021-04-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Drep-HIV-PT1 0.2mg and CN54gp140/MPLA-L (Experimental): 0.1mL of DREP-HIV-PT1 will be diluted with saline (Sodium Chloride for Injection, 0.9%) and administered intramuscularly (total volume of 0.5mL) in the LEFT deltoid muscle using a needle-free device (Pharmajet Stratis®)
  0.4mL of MPLA-L from a vial containing 0.55mL of MPLA-L (25µg/mL) and add this to a vial containing 0.35mL of CN54gp140 (500µg/mL). The vial contents will be mixed by gentle agitation and 0.45mL of will be withdrawn from the vial to make a concentration of 100µg CN54gp140 and 5µg MPLA-L . The combined products will be injected into the RIGHT deltoid muscle using a needle and syringe.
  Interventions: Biological: Drep-HIV-PT1 0.2mg and CN54gp140/MPLA-L
- Drep-HIV-PT1 1.0mg and CN54gp140/MPLA-L (Experimental): 0.5mL of DREP-HIV-PT1 will be administered intramuscularly in the LEFT deltoid muscle using the a needle-free device (Pharmajet Stratis®)
  0.4mL of MPLA-L from a vial containing 0.55mL of MPLA-L (25µg/mL) and add this to a vial containing 0.35mL of CN54gp140 (500µg/mL). The vial contents will be mixed by gentle agitation and 0.45mL of will be withdrawn from the vial to make a concentration of 100µg CN54gp140 and 5µg MPLA-L . The combined products will be injected into the RIGHT deltoid muscle using a needle and syringe.
  Interventions: Biological: DREP-HIV-PT1 1mg and CN54gp140/MPLA-L (see above)
- DNA HIV PT123 4mg and CN54gp140/MPLA-L (Experimental): 1ml of DNA-HIV-PT123 will be injected into the LEFT deltoid muscle using a needle and syringe.
  0.4mL of MPLA-L from a vial containing 0.55mL of MPLA-L (25µg/mL) and add this to a vial containing 0.35mL of CN54gp140 (500µg/mL). The vial contents will be mixed by gentle agitation and 0.45mL of will be withdrawn from the vial to make a concentration of 100µg CN54gp140 and 5µg MPLA-L . The combined products will be injected into the RIGHT deltoid muscle using a needle and syringe.
  Interventions: Biological: DNA-HIV-PT123 4mg and CN54gp140/MPLA-L

INTERVENTIONS:
Biological: Drep-HIV-PT1 0.2mg and CN54gp140/MPLA-L — 1. Drep-HIV-PT1 The DREP-HIV-PT1 is a vaccine designed to elicit an immune response against human immunodeficiency virus-1 (HIV-1) and prevent infection by HIV-1 and/or disease caused by HIV-1. It is an alphavirus-based DNA replicon in which the sequences coding for the viral capsid and envelope have been replaced by the sequences encoding HIV-1 gp140 (96ZM651) antigen.
  2. CN54gp140+MPLA-L. Recombinant CN54gp140 is a HIV-1 envelope protein from the clade C strain 97/CN/54 isolate, which comprises a sequence of 634 amino acids. MPLA is a non-toxic version of LipoPolySaccharide (LPS), which is isolated from the LPS lipid A region of Salmonella Minnesota R595 and retains the immune-stimulatory properties of LPS, but exhibits low toxicity.
  Arms: Drep-HIV-PT1 0.2mg and CN54gp140/MPLA-L
Biological: DREP-HIV-PT1 1mg and CN54gp140/MPLA-L (see above) — 1. Drep-HIV-PT1 1mg (see above)
  2. Drep-HIV-PT1 1mg (see above)
  Arms: Drep-HIV-PT1 1.0mg and CN54gp140/MPLA-L
Biological: DNA-HIV-PT123 4mg and CN54gp140/MPLA-L — 1. DNA-HIV-PT123 HIV vaccine includes three DNA plasmids that encode clade C ZM96 Gag, clade C ZM96 Env, and CN54 Pol-Nef
  2. CN54gp140/MPLA-L Recombinant CN54gp140 is a HIV-1 envelope protein from the clade C strain 97/CN/54 isolate, which comprises a sequence of 634 amino acids. MPLA is a non-toxic version of LipoPolySaccharide (LPS), which is isolated from the LPS lipid A region of Salmonella Minnesota R595 and retains the immune-stimulatory properties of LPS, but exhibits low toxicity.
  Arms: DNA HIV PT123 4mg and CN54gp140/MPLA-L

SUMMARY:
EHVA P01 is an international, phase I, prophylactic HIV vaccine trial to evaluate the safety and immunogenicity of HIV Clade C DREP alone and in Combination with a Clade C ENV protein in healthy HIV-uninfected adults.

DETAILED DESCRIPTION:
The study is looking at the use of a new vaccine against the HIV virus. There are two parts to the study. One part is open-label to assess the safety of this vaccine, since this will be the first time that it has been used in humans. The second part is to see how well, and for how long, the vaccine activates the immune system. But this trial is not looking at whether or not the vaccine is effective in terms of protection against HIV. It is just assessing whether and how well the immune system responds.

Since this is the first time the vaccine has been used in humans, the safety will be assessed initially in healthy young adults. 10 participants aged 18-55 years will be given one of two different doses (0.2 and 1.0 mg) by injection into the arm muscle. There will be careful monitoring for any reactions to the vaccine.

As long as there are no safety concerns, the second part of the study can then be started. This will see how well the immune system has been activated using different dose levels of the vaccine. About 60 participants aged 18-55 years will be given one of three doses schedules (0.2mg, 1.0mg of the new vaccine and 4.0mg of a conventional vaccine). Chance will determine which dose each individual is given. Participants are only blind to the dose of vaccine administered but laboratory technicians assessing the safety parameters and immune responses will be blinded. The vaccine is given by injection into the muscle of the upper arm. Two injections, four weeks apart, are needed for the first part of the trial. There are three vaccinations in part two of the trial. There are likely to be mild side-effects near to the injection site. There may also be more general side-effects such as headache, temperature and chills. Participants will be asked to record any symptoms in an online diary. In order to see how well the immune system is responding, participants will need to give blood samples at several time points. The vaccines are not made from HIV and cannot cause HIV infection. However, the vaccines are likely to cause participants to produce antibodies against HIV that are detected by the rapid HIV antibody tests that are used in routine testing and a test that detects and measures antibodies in the blood used for confirmation. It is recommended that participants have an up to date vaccination status for any required immunisations including authorised COVID-19 vaccines. Vaccination with licensed (including authorised COVID-19) vaccines should be avoided from 28 days before and after each injection .

An independent steering committee will regularly review the information on safety and look at the immune responses to see which dose of the candidate vaccine could go forward to effectiveness testing in future trials. Before this study can start, the protocol describing the procedures and information to be provided to volunteers will be reviewed by the national drug authority and a multi-centre research ethics committee in the participating countries.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18- 55 years on the day of screening
2. BMI between 18-30 kg/m2 (inclusive)
3. Unlikely to acquire HIV during follow-up
4. Willing and able to provide written informed consent
5. If female and of childbearing potential* age and not sterilised, willing to use a highly effective method of contraception from screening until 12 weeks after last injection
6. If male and not sterilised, willing to avoid impregnating female partners from screening until 12 weeks after last injection**
7. Willing to avoid all other vaccines from 28 days before the first injection through to 28 days after subsequent study injections
8. Willing and able to comply with visit schedule and provide blood samples
9. Being covered by medical insurance or in National Healthcare System

   * A woman will be considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

     * It is recommended that participants have an up to date vaccination status for any required immunisations including authorised COVID-19 vaccines

Exclusion Criteria:

1. Pregnant or lactating
2. Has a significant clinical history, physical finding on clinical examination during screening, or presence of a disease that is active or requires treatment to control it, including cardiac, respiratory, endocrine, metabolic, autoimmune, liver, neurological, oncological, psychiatric, immunosuppresive/immunodeficient or other disorders which in the opinion of the investigator is not compatible with healthy status, may compromise the volunteer's safety, preclude vaccination or compromise interpretation of the immune response to vaccine. Individuals with mild/moderate, well-controlled comorbidities are allowed.
3. HIV 1 or 2 infection or indeterminate test at screening
4. History of anaphylaxis or angioedema
5. History of severe or multiple allergies to drugs or pharmaceutical agents
6. Known hypersensitivity to any component of the vaccine formulation used in this trial
7. History of severe local or general reaction to vaccination defined as

   1. local: extensive, indurated redness and swelling involving most of the arm, not resolving within 72 hours
   2. general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
8. Receipt of any experimental vaccine within 5 years from screening.
9. Receipt of blood products or immunoglobulins within 18 weeks of screening.
10. Receipt any of immunosuppressive agents within 18 weeks of screening by any route other than skin and intranasal.
11. Detection of antibodies to hepatitis B & C
12. Participating in another clinical trial with an investigational drug or device, or treated with an investigational drug within 28 days of screening
13. Any of the values that are confirmed on repeat testing as defined in protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Part 1- Dose Escalation- Any adverse reaction that results in a clinical decision to stop immunisations | From week 0 up to Week 4
  Any adverse reaction that results in a clinical decision that no further immunisations can be given
Part 2- Randomised Comparison - Any adverse reaction that results in a clinical decision to stop immunisations | From week 0 up to Week 9
  Any adverse reaction that results in a clinical decision that no further immunisations can be given
PART 2 Randomised comparison- Total IgG Binding antibody response rate | At week 26
  1. Env-specific total IgG binding antibody response rates assessed by binding antibody multiplex assay (BAMA)
  2. Magnitude of Env-specific total IgG binding antibody responses to HIV-1 Env proteins assessed by binding antibody multiplex assay (BAMA)

SECONDARY OUTCOMES:
Part 1- Dose Escalation - Occurrence of Adverse events | From week 0 to Week 11
  1. Grade 3 or worse local or systemic solicited adverse events
  2. Grade 1 or 2 local or systemic solicited adverse events
  3. Non-solicited adverse events
  4. Serious adverse events
Part 1- Dose Escalation - Binding antibodies to ZM96gp140 | At week 6 and Week 26
  Binding antibodies to ZM96gp140 measured by ELISA
PART 2 Randomised comparison- Total IgG binding antibody response rates | 1, 2 (At week 6); 3,5 (At week 26) and 4,6 (At week 36)
  1. Env-specific total IgG binding antibody response rates assessed by binding antibody multiplex assay (BAMA)
  2. Magnitude of Env-specific total IgG binding antibody responses to HIV-1 Env proteins assessed by binding antibody multiplex assay (BAMA)
  3. Breadth of Env-specific total IgG binding antibody responses to HIV-1 Env proteins assessed by binding antibody multiplex assay (BAMA)
  4. Durability of Env-specific total IgG binding antibody responses to HIV-1 Env proteins assessed by binding antibody multiplex assay (BAMA)
  5. Response rate and magnitude of Env-specific CD4+ and CD8+ T-cell responses measured by intracellular cytokine staining (ICS)
  6. Durability of Env-specific CD4+ and CD8+ T-cell responses measured by intracellular cytokine staining

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - CIC Cochin, Paris, Paris Cedex 14
  - Hôpital Henri Mondor, Créteil, Paris
- CHUV, Lausanne, Canton of Vaud, Switzerland
- Chelsea and Westminster Hospital, London, United Kingdom